CLINICAL TRIAL: NCT01091883
Title: Phase IIIA Study Comparing the Safety and Effectiveness of MR Guided Focused Ultrasound and External Beam Radiation for Treatment of Metastatic Bone Tumors and Multiple Myeloma
Brief Title: Study Comparing the Safety and Effectiveness of Magnetic Resonance Guided Focused Ultrasound (MRgFUS) and External Beam Radiation (EBRT) for Treatment of Metastatic Bone Tumors and Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BM016
Record Dates: First submitted 2010-03-18; First posted 2010-03-24 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Bone Cancer; Bone Metastases; Pain
Keywords: Bone cancer; Bone Metastases; pain palliation; metastasis; breast cancer; lung cancer; prostate cancer; cancer related pain; tumors
MeSH Terms: conditions — Bone Neoplasms; Pain; Neoplasm Metastasis; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Cancer Pain; Neoplasms | interventions — Radiation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exablate treatment (Experimental): Exablate 2000
  Interventions: Device: Exablate treatment
- Radiation (Active Comparator): External Beam Radiation
  Interventions: Radiation: Radiation

INTERVENTIONS:
Device: Exablate treatment — MR Guided Focused Ultrasound
  Arms: Exablate treatment
Radiation: Radiation — External Beam Radiation
  Arms: Radiation

SUMMARY:
The goal of this study is to collect comparative data on safety and efficacy of MR Guided Focused Ultrasound and External Beam Radiation for treatment of metastatic bone tumors or multiple myeloma.

DETAILED DESCRIPTION:
Bone is the third most common organ involved by metastatic disease behind lung and liver [6]. In breast cancer, bone is the second most common site of metastatic spread, and 90% of patients dying of breast cancer have bone metastasis. Breast and prostate cancer metastasize to bone most frequently, which reflects the high incidence of both these tumors, as well as their prolonged clinical courses. Post-cancer survival has increased with improvement in early detection and treatments. As a consequence, the number of patients developing metastatic bone disease during their lifetime has also increased.

Current treatments for patients with bone metastases are primarily palliative and include localized therapies (radiation and surgery), systemic therapies (chemotherapy, hormonal therapy, radiopharmaceutical, and bisphosphonates although the primary goal of the use of these therapies are often to address the disease itself), and analgesics (opioids and non-steroidal anti-inflammatory drugs). Recently, radiofrequency ablation has been tested as a treatment option for bone metastases [8]. Currently, an off label use of Cryoablation techniques are being tested as another alternative for bone Mets palliation. The main goals of these treatments are improvement of quality of life and functional level. These goals can be further described:

* Pain relief
* Preservation and restoration of function
* Local tumor control
* Skeletal stabilization

Treatment with external beam radiation therapy (EBRT) is the standard of care for patients with localized bone pain, and results in the palliation of pain for many of these patients. Twenty to 30% of patients treated with radiation therapy do not experience pain relief [9-13]. Re-treatment rates are generally reported in the range of 10-25%. Many patients with relapsed pain or poor response to initial radiation may be lost to follow up or may not be referred back to oncologists for consideration of re-radiation. In addition to relapse and re-treatment, there is an increased risk of pathologic fracture in the peri-radiation period. The fracture rate reported in radiation studies is generally in the range of 1% to 8%. The hyperemic response weakens the adjacent bone and increases the risk of spontaneous fracture. Furthermore, patients who have recurrent pain at a site previously irradiated may not be eligible for further radiation therapy secondary to limitations in normal tissue tolerance. Hesitation on the part of physicians to use a larger dose may be related to increased long-term toxicity. Larger radiation dose produces a greater risk of complications such as fibrosis of normal soft tissue, which can cause a decrement in the quality of life in cases of life expectancy longer than 6 months. There may also be a greater incidence of acute side effects of nausea and vomiting if the treatment field includes the stomach. The percent of patients experiencing vomiting following EBRT ranges from about 5% to 30%.

A palliative treatment for painful bone metastases that is non-invasive, without long-term toxicity and having minimal complications would be a useful tool for treating physicians and also a beneficial option for patients suffering from painful bone metastases. Results of preliminary studies indicate that ExAblate treatment of painful bone metastases may be a beneficial treatment option [14, 15]. The ExAblate system is a non-invasive thermal ablation device used in the coagulation of various types of soft tissue. The ExAblate system has the potential to achieve the first three of the four previously mentioned goals in the treatment of bone tumors; namely pain relief, preservation and restoration of functional levels and local tumor control [11].

This study will compare the safety and effectiveness of MR Guided Focused Ultrasound and External Beam Radiation for treatment of metastatic bone tumors or multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18 years and older.
2. Able and willing to give consent and to attend all study visits
3. Patients with bone metastasis or primary bone lesion identifiable by imaging techniques.
4. Worst NRS Pain Score of ≥ 4 from the tumor to be treated.
5. Targeted tumor(s) are accessible to both ExAblate and EBRT (ExAblate accessible lesions are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3 - L5), Sacral vertebra (S1 - S5), please see ExAblate "Information for Prescribers".
6. Targeted tumor(s) area is smaller than 100cm2.
7. Tumor(s) clearly visible by non-contrast MRI.
8. No radiation therapy to the treated lesion during one month prior to enrollment.
9. Radiation therapy is not contraindicated
10. Bisphosphonate, chemo or hormone therapy intake should remain stable throughout follow up duration.

Exclusion Criteria:

1. Patients who either

   * Need pre-treatment surgical stabilization of the affected bony structure OR
   * prior surgical stabilization of tumor site
2. Targeted tumor is in a vertebra body or in the posterior aspects of the cervical part of the vertebral column.
3. Targeted tumor is in the skull.
4. Patients on anti-coagulation therapy or with an underlying uncontrolled bleeding disorder.
5. Patients with life expectancy < 6-Months.
6. Patients with unstable cardiac status including:

   * Unstable angina pectoris on medication.
   * Patients with documented myocardial infarction within last 40 days to protocol entry.
   * Congestive heart failure NYHA Class IV
7. Severe hypertension (diastolic BP > 100 on medication).
8. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted ferromagnetic objects/devices.
9. Known intolerance or allergies to MRI contrast agent (e.g. Gadolinium or Magnevist)
10. KPS score of below 60
11. Severe cerebro-vascular disease (multiple CVA or CVA within 6 months)
12. Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hrs.)
13. Target tumor is less then 1cm from spinal cord, skin, or hollow viscera.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Safety of treatment | 6 months
  Incidence and severity of adverse events associated with the ExAblate MRgFUS bone system used in the palliation of pain due to metastatic bone tumors or multiple myeloma to that of EBRT
NRS score | 6 months
  Effect of treatment with MRgFUS ExAblate Bone System (BS) of painful bone tumors or multiple myeloma

SECONDARY OUTCOMES:
Pain Medication dose and quantity | 6 months
  Decrease in analgesics/opiate
Quality of Life score | 6 months
  Improved quality of life (measured by questionnaires)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei City, Taipei, Taiwan

REFERENCES:
- [Derived] Bertrand AS, Iannessi A, Natale R, Beaumont H, Patriti S, Xiong-Ying J, Baudin G, Thyss A. Focused ultrasound for the treatment of bone metastases: effectiveness and feasibility. J Ther Ultrasound. 2018 Nov 30;6:8. doi: 10.1186/s40349-018-0117-3. eCollection 2018. PMID 30519467
- See also: Sponsor's Website — http://www.insightec.com